CLINICAL TRIAL: NCT05417321
Title: A Phase I/II, Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of HB0036 in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety and Efficacy of HB0036 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB0036-01
Record Dates: First submitted 2022-05-30; First posted 2022-06-14 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor; NSCLC

STUDY DESIGN:
Intervention Model Description: A single-subject cohort will be enrolled at the protocol starting dose of HB0036 every 3 weeks (Q3W). Dose escalation will proceed to the next main dose level according to the 3+3 dose-escalation procedure until the MTD/OBD is reached. Phase II of the study will be initiated at the Sponsor's discretion at the dose level and treatment schedule which was established as the recommended Phase 2 dose (RP2D) in the dose-escalation phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB0036 (Experimental): HB0036 IV every 3 weeks (q3w)
  Interventions: Drug: HB0036

INTERVENTIONS:
Drug: HB0036 — Patients will be assigned to dose regimens in the order of enrollment, and they will receive their assigned fixed dose of HB0036 via intravenous infusion. HB0036 IV every 3 weeks (q3w).
  Other Names: Anti-PD-L1 and anti-TIGIT bifunctional molecule

SUMMARY:
It is a Phase I/II, Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of HB0036 in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a phase Ⅰ/Ⅱ, multicenter, open-label, first-in-human study in patients with advanced solid tumors. During the phase Ⅰ study, the safety and tolerability of HB0036 will be evaluated in patients with advanced solid tumors. In the phase Ⅱ study, the safety and efficacy of HB0036 at the RP2D will be evaluated in cohorts of patients with NSCLC and/or other solid tumors.

A Safety Review Committee (SRC) will be established throughout the study period, consisting of the principal investigator, representatives of the contract research organization (CRO) (medical inspectors and other relevant personnel), and the Sponsor's medical monitor. The SRC will evaluate safety data based on the study process. The SRC may recommend extended doses, possible changes in the frequency of administration, and extended tumor types for safety reasons based on existing studies prior to starting the phase II study.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the following criteria to be eligible for participation in this study:

1. Male or female. Age ≥ 18 years;
2. Phase I: Patients with histologically or cytologically confirmed locally advanced, recurrent, or metastatic solid tumors (or clinically diagnosed hepatocellular carcinoma) that failed all standard therapies known to provide clinical benefit; [These solid tumors include but not limit to: non-small cell lung cancer, esophageal squamous cell carcinoma, melanoma, head and neck squamous cell carcinomas, hepatocellular carcinoma, gastric or gastroesophageal junction adenocarcinoma, renal cell carcinoma, etc.];
3. Phase II: Histologically or cytologically documented locally advanced, recurrent or metastatic cancer. There will be several tumor-specific cohorts Advanced non-small cell lung cancer cohort Histologically or cytologically documented locally advanced, recurrent or metastatic NSCLC; Confirmed availability of representative tumor specimens in formalin-fixed paraffin-embedded (FFPE）blocks or at least 5 stained serial slides or fresh biopsied specimens (preferred),samples obtained before adjuvant / neoadjuvant chemotherapy are allowed only if biopsy cannot be performed; Tumor PD-L1 expression with a TPS≥1 %; Negative for actionable molecular markers [including but not limited to: epidermal growth factor receptor (EGFR) mutations, anaplastic lymphoma kinase (ALK) gene fusion mutation, etc.]； Assessed by the investigator as likely to benefit from the study drug therapy; and should have progressed at least one prior systemic therapy regimen.

   Advanced other cancer cohort Histologically or cytologically documented locally advanced, recurrent or metastatic cancer (esophageal squamous cell carcinoma, melanoma) Other tumor histologies will be evaluated pending data from the dose escalation phase that may inform on possible efficacy in select tumors
4. At least one measurable lesion( assessable lesion only accepted during accelerated titration stage) as per RECIST v. 1.1 defined as non-nodal lesions having at least one dimension with a minimum size of 10 mm in the longest diameter by CT or MRI scan or ≥15 mm in short axis for nodal lesions. Radiographic disease assessment at baseline can be performed up to 21 days prior to the first dose.

   Note: Tumour lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
6. Life expectancy ≥12 weeks
7. Adequate organ function within 14 days of the first dose as defined by the following criteria:

   a) Hematology
   * absolute neutrophil count (ANC) ≥ 1.5×109/L;

     ② platelets (PLT) ≥ 75×109/L;

     ③ hemoglobin (HGB) ≥ 90 g/L; Note: The above three items require that patients should not have received any blood component or cell growth factor supportive therapy within two weeks prior to blood sampling.

     b) Renal function: Calculated creatinine clearance (CrCL) > 50 mL/min (Cockroft-Gault Equation); c) Liver function:
   * AST and ALT ≤ 2.5×ULN; AST or ALT ≤5×ULN if liver metastases are present;

     ② Total bilirubin (TBIL) ≤ 1.5×ULN; ≤3 X ULN for patients with Gilbert's disease; d) Coagulation function:
   * International normalized ratio (INR)or prothrombin time (PT)≤ 1.5×ULN (unless patient on oral anticoagulant with stable dose); ② Activated partial thromboplastin time (APTT)≤ 1.5×ULN;
8. Women of childbearing potential must confirm a negative serum or urine pregnancy test within 3 days prior to the initiation of study treatment; Fertile patients and their partners must agree to use effective contraceptives for the duration of study drug use and for 90 days after the last administration of study treatment
9. Recovery to Grade 0-1 from adverse events (AEs) related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, and endocrinopathies controlled with hormone replacement therapy
10. The subject is able to understand and willing to sign the ICF; willing and able to comply with all study procedures.

Exclusion Criteria

Patients are excluded from the study if any of the following criteria apply:

1. Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma. Patients with prostate cancer that is under active surveillance are eligible.
2. Phase I: Patients may have received single agent treatments targeting the TIGIT pathway.

   Phase II: Have received previous simultaneous therapy with a PD-1 pathway inhibitor and a TIGIT inhibitor; previous monotherapy with TIGIT/PD-1/PD-L1 inhibitor is allowed.
3. Have received antibiotics lasting over 1 week within 28 days prior to first dose;
4. Have clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously-treated brain or meningeal metastases may participate and be eligible for treatment provided they are stable and asymptomatic. Patients with asymptomatic brain metastasis or subjects who are symptomatically stable after treatment and are on < 10 mg/d prednisone or equivalent are eligible.
5. Have history of interstitial lung disease or non-infectious pneumonitis (except from radiotherapy);
6. Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
7. History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for grade 3 endocrinopathy that is managed with hormone replacement therapy).
8. Use of systemic corticosteroids in a dose equivalent to >10 mg/day of prednisone or other immunosuppressive agent < 2 weeks prior to screening; the use of topical, intraocular, intraarticular, intranasal, or inhaled corticosteroids and systemic steroids to prevent (e.g., allergy to contrast agents) or treat non-autoimmune condition (e.g., delayed hypersensitivity caused by exposure to allergens) or short course (< 5 days) will be allowed
9. Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study entry; palliative radiotherapy to a single area < 2 weeks prior to study screening is permitted. Measurable lesions cannot be previously irradiated unless they have demonstrated growth after radiation therapy (RT).
10. Major surgery (except for diagnostic needle biopsy or intravenous catheterization) or chemotherapy/ interventional therapy/radiation therapy/ablation therapy < 4 weeks prior to the first dose;
11. Cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure < 6 months of study entry; mean ECG QT-interval corrected according to Fridericia's formula (QTcF) > 470 milliseconds (ms) obtained from three ECGs; uncontrolled arrhythmia < 3 months of study entry. Patients with rate-controlled arrhythmias may be eligible for study entry at discretion of the Investigator.
12. Patients who have previously received allogeneic stem cell or solid organ transplantation.
13. Have received or will receive a live vaccine within 4 weeks prior to the first dose, except COVID-19 vaccine.
14. Patients whose existing significant clinical abnormalities or laboratory abnormalities may affect the evaluation of the study drug by the Investigator's judgement, e.g. uncontrolled active infection (>Grade 2, CTCAE v5.0), uncontrolled diabetes, poorly controlled hypertension with the combination of the two drugs (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), congestive heart failure, myocardial infarction within 24 weeks, etc.;.
15. Positive results for HIV test.
16. Active hepatitis B or C. Patients with asymptomatic hepatitis B virus carriers (HBV DNA titer < 1000 CPS /mL or 200 IU/mL) or cured hepatitis C (negative HCV RNA test) may be enrolled;
17. Positive COVID-19 qRT-PCR or rapid screening test during screening; can be eligible after quarantine (14 days) if COVID-19 test becomes negative.
18. Patients with active tuberculosis (TB) who are receiving anti-TB treatment or who received anti-TB treatment within 1 year prior to screening;
19. Women who are pregnant or lactating, or women of childbearing potential who do not wish to use effective contraception method during the trial.
20. Men with a partner of childbearing potential who do not consent to use acceptable methods of birth control during treatment and for an additional 90 days after the last administration of study drug.
21. History of severe allergic reactions, grade 3-4 allergic reactions to treatment with another monoclonal antibody, or known to be allergic to protein drugs or recombinant proteins or excipients in HB0036 drug formulation;
22. Patients who have participated in any clinical trial of a drug or medical device within 4 weeks prior to the first dose.
23. Abuse of alcohol, cannabis- derived products or other drugs; can be eligible with remote history of abuse more than 2 years.
24. Any other serious underlying medical condition (e.g., active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, cardiac conditions), or psychiatric, psychological, familial condition or geographical location that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment.
25. Other conditions which would make it inappropriate for the patient to participate as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 12 Months
  Number of participants with a Dose Limiting Toxicity (DLT) [ Time Frame: During the first 21 days ]DLTs will be assessed during the first 21 days of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected or definite relationship to study drug.
MTD | Up to 24 Months
  MTD or OBD and/or RP2D.

SECONDARY OUTCOMES:
AUC | Up to 24 Months
  Area Under concentration-time Curve (AUC)
Cmax | Up to 24 Months
  Maximum serum concentration (Cmax)
Tmax | Up to 24 Months
  half-life time of maximum concentration

OTHER OUTCOMES:
ORR assessment in dose-escalation phase | Up to 24 Months
  Overall response rate (ORR) as measured by RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, MD/PHD, Study Director — Shanghai Huaota Biopharmaceutical Co., Ltd.
Locations (4):
- United States (3):
  - Horizon Oncology, Lafayette, Indiana
  - Next Oncology, San Antonio, Texas
  - Summit Cancer Centers, Spokane, Washington
- Shandong Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No